CLINICAL TRIAL: NCT05891665
Title: The Effectiveness of Minimally-invasive Corticotomy-assisted Orthodontic Treatment of Palatally Impacted Canines in Terms of Treatment Duration and Dentoalveolar Changes Compared to the Traditional Method: A Randomized Controlled Trial.
Brief Title: Evaluation of the Accelerated Traction of Impacted Canines in Terms of Speed and Changes in the Dental Arches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-10-2023
Record Dates: First submitted 2023-05-14; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Impacted Tooth With Abnormal Positioning
Keywords: Canine impaction; Acceleration of tooth movement; Corticotomy; Minimally invasive acceleration; Maxillary canine impaction; Withdrawal of an impacted canine; Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with the acceleration method (Experimental): Patients will be treated using fixed orthodontic appliances assisted by minimally-invasive corticotomy (osteoperforations and piezocision) to accelerate impacted canines' traction after levelling and aligning the upper dental arch and opening an appropriate distance.
  Interventions: Procedure: Corticotomy
- Patients treated with the traditional traction technique (Active Comparator): Patients will be treated using the fixed orthodontic appliances to track the palatally impacted canines after levelling and aligning the upper dental arch and opening an appropriate space to receive the impacted canine.
  Interventions: Procedure: Traditional traction of the impacted canine without corticotomy

INTERVENTIONS:
Procedure: Corticotomy — A corticotomy procedure will be applied with some osteoperforations during the surgical exposure of the impacted canine. Then this will be followed after 8 weeks with another surgical stimulation using piezosurgery.
  Arms: Patients treated with the acceleration method
Procedure: Traditional traction of the impacted canine without corticotomy — In this group of patients, the traction of the impacted canine will be performed traditionally without the involvement of additional surgical intervention.
  Arms: Patients treated with the traditional traction technique

SUMMARY:
The time required for orthodontic traction of impacted canines after surgical exposure is a particularly troubling clinical problem because it prolongs the orthodontic treatment duration. During traction process, several complications could result in alveolar bone loss, root resorption of the adjacent teeth, ankylosis, discoloration, loss or vitality and gingival recession. Accordingly, and due to the lack of studies concerned with accelerating the traction movement of the impacted canines, we conducted this study to evaluate the effectiveness of some surgical interventions (corticotomy and Piezocision) in increasing the rate of orthodontic traction movement. We also aimed to evaluate dentoalveolar changes associated with the use of such accelerating procedures compared with the conventional traction method.

DETAILED DESCRIPTION:
Adult patients with unilateral palatally impacted canines will be included in this study. One of patient groups will be treated using fixed orthodontic appliances in combination with some accelerated surgical interventions, while the second patient group will be treated using the traditional treatment method. The velocity of traction movement will be assessed in the two groups. The differences between the two groups in terms of the total treatment duration and the traction duration will be evaluated.

Dentoalveolar changes associated with the use of such accelerating procedures will be assessed by several variables studied on cone-beam computed tomography (CBCT) images. In this study, two groups are going to be evaluated: (1) patients treated in the traditional manner, (2) patients will undergo corticotomy-assisted traction of the impacted canines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 28.
2. Unilateral palatally or mid-alveolar upper impacted canine.
3. The impacted canine crown not exceeding the middle of the lateral incisor root.
4. Absence of root resorption of the lateral incisors.
5. No contact between the canine crown and the lateral incisor root.
6. Individuals not previously receiving orthodontic treatment.
7. No use of any medications that may affect the orthodontic movement.

Exclusion Criteria:

1. Bilateral or buccal canine impaction cases.
2. More than 45-degree angle between the canine's longitudinal axis and the vertical facial plane.
3. Any medical condition that prevents oral surgery.
4. Oral structural abnormality that is inherited or congenital.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Traction time | At the end of the traction stage which is expected to happen within 6 to 8 months
  The interval between the onset of orthodontic traction on the impacted canine and the emergence of half of its clinical crown.
Total treatment time | At the end of the orthodontic treatment which is expected to happen between 15 to 24 months.
  The time between the bonding of the fixed orthodontic appliance until it is removed.
Velocity of the traction movement | At the end of the traction stage which is expected to happen within 6 to 8 months
  Calculated by dividing the depth of impaction, which defined as the distance from the impacted canine cusp tip to the occlusal plane, by the traction duration

SECONDARY OUTCOMES:
Bone support ratio of the aligned canine | At the end of the orthodontic treatment which is expected to happen between 15 to 24 months.
  Alveolar bone height is the distance from the root apex of the canine to the alveolar crest (measured in mm), and canine root length is the distance from the root apex of the canine to the midpoint of a line connecting the mesial and distal points on the cementoenamel junction (measured in mm). The ratio will be calculated by dividing the alveolar bone height by the canine root length.
Bone support ratio of the contralateral naturally erupting canine | At the end of the orthodontic treatment which is expected to happen between 15 to 24 months.
  Alveolar bone height is the distance from the root apex of the naturally erupting canine to the alveolar crest (measured in mm), and canine root length is the distance from the root apex of the naturally erupting canine to the midpoint of a line connecting the mesial and distal points on the cementoenamel junction (measured in mm). The ratio will be calculated by dividing the alveolar bone height by the canine root length.
Bone support ratio of the adjacent lateral incisor | At the end of the orthodontic treatment which is expected to happen between 15 to 24 months.
  Alveolar bone height is the distance from the root apex of the adjacent lateral incisor to the alveolar crest (measured in mm), and the lateral incisor's root length is the distance from the root apex of the lateral incisor to the midpoint of a line connecting the mesial and distal points on the cementoenamel junction (measured in mm). The ratio will be calculated by dividing the alveolar bone height by the lateral incisor's root length.
Bone support ratio of the adjacent first premolar | At the end of the orthodontic treatment which is expected to happen between 15 to 24 months.
  Alveolar bone height is the distance from the root apex of the adjacent first premolar to the alveolar crest (measured in mm), and the first premolar's root length is the distance from the root apex of the first premolar to the midpoint of a line connecting the mesial and distal points on the cementoenamel junction (measured in mm). The ratio will be calculated by dividing the alveolar bone height by the first premolar root length.
Change of the root length of the adjacent lateral incisor | (1) The first assessment time is at one day before the beginning of orthodontic treatment and the (2) second assessment time is at one week following the end of the orthodontic treatment
  Resorption of adjacent lateral root will be evaluated by comparing the root length before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mahran R. Mousa, DDS MSc, Principal Investigator — PhD student at the Department of Orthodontics; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Professor of Orthodontics, Faculty of Dentistry, University of Damascus; Omar Heshmeh, DDS MSc PhD, Study Chair — Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry, University of Damascus
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Ibrahim HM, Hajeer MY, Alkhouri I, Zinah E. Leveling and alignment time and the periodontal status in patients with severe upper crowding treated by corticotomy-assisted self-ligating brackets in comparison with conventional or self-ligating brackets only: a 3-arm randomized controlled clinical trial. J World Fed Orthod. 2022 Feb;11(1):3-11. doi: 10.1016/j.ejwf.2021.09.002. Epub 2021 Oct 21. PMID 34688577
- [Background] Becker A, Chaushu S. Success rate and duration of orthodontic treatment for adult patients with palatally impacted maxillary canines. Am J Orthod Dentofacial Orthop. 2003 Nov;124(5):509-14. doi: 10.1016/s0889-5406(03)00578-x. PMID 14614417
- [Background] Becker A, Kohavi D, Zilberman Y. Periodontal status following the alignment of palatally impacted canine teeth. Am J Orthod. 1983 Oct;84(4):332-6. doi: 10.1016/s0002-9416(83)90349-4. PMID 6578683
- [Background] Smailiene D, Kavaliauskiene A, Pacauskiene I, Zasciurinskiene E, Bjerklin K. Palatally impacted maxillary canines: choice of surgical-orthodontic treatment method does not influence post-treatment periodontal status. A controlled prospective study. Eur J Orthod. 2013 Dec;35(6):803-10. doi: 10.1093/ejo/cjs102. Epub 2013 Jan 24. PMID 23349422
- [Background] Fischer TJ. Orthodontic treatment acceleration with corticotomy-assisted exposure of palatally impacted canines. Angle Orthod. 2007 May;77(3):417-20. doi: 10.2319/0003-3219(2007)077[0417:OTAWCE]2.0.CO;2. PMID 17465647
- [Background] Mousa MR, Hajeer MY, Burhan AS, Heshmeh O. The Effectiveness of Conventional and Accelerated Methods of Orthodontic Traction and Alignment of Palatally Impacted Canines in Terms of Treatment Time, Velocity of Tooth Movement, Periodontal, and Patient-Reported Outcomes: A Systematic Review. Cureus. 2022 May 10;14(5):e24888. doi: 10.7759/cureus.24888. eCollection 2022 May. PMID 35572459
- [Background] Parkin NA, Almutairi S, Benson PE. Surgical exposure and orthodontic alignment of palatally displaced canines: can we shorten treatment time? J Orthod. 2019 Jun;46(1_suppl):54-59. doi: 10.1177/1465312519841384. Epub 2019 Apr 1. PMID 31056030